CLINICAL TRIAL: NCT06405477
Title: EFFECTS OF L-ARGININE SUPPLEMENTATION ON THE RECOVERY OF CARDIORESPIRATORY PARAMETERS AFTER SUBMAXIMAL EXERCISE TEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Luana Almeida Gonzaga, Principal investigator, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LargExBr
Record Dates: First submitted 2024-04-26; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Nutrition, Healthy
MeSH Terms: interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sun (Experimental): We are blind and don't know which group is which.
  Interventions: Dietary Supplement: L-arginine; Dietary Supplement: Placebo
- Moon (Placebo Comparator): We are blind and don't know which group is which.
  Interventions: Dietary Supplement: L-arginine; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-arginine — Capsules of 3 grams of L-arginine per Dose
Dietary Supplement: Placebo — Capsules of 3 grams of maize Starch per Dose

SUMMARY:
L-Arginine is an amino acid capable of stimulating the production of nitric oxide (NO) metabolites. NO is responsible for several important activities of the body, such as: helping to regulate vasodilation, blood flow, mitochondrial respiration, platelet function and increasing growth hormone levels, but the effects on the recovery of cardiorespiratory parameters after exercise testing maximum need to be clarified.

DETAILED DESCRIPTION:
The protocols will be carried out at the Stress Physiology Laboratory of the Faculty of Science and Technology, UNESP-Presidente Prudente. The execution time of the protocols will be between 5:00 pm and 9:00 pm, to standardize the circadian influence on the evaluated parameters, the environmental climate will be controlled with a temperature between 23ºC and 24 ºC and humidity between 60% and 70%. Volunteers will be instructed not to drink alcoholic or caffeine-based drinks for 12 hours before all protocols, to consume a light meal and 500 ml of water two hours before and to avoid vigorous physical exertion the day before. The experimental procedure will be divided into two stages, all carried out on a treadmill, with a minimum interval of 48 hours between them, in order to allow adequate recovery. Before the start of the first stage of the protocols, anthropometric measurements will be taken, body weight using a digital scale and height using a stadiometer.

Before the beginning of each stage, a Polar RS800CX heart rate monitor will be placed to record the heart rate (HR) and its variability, remaining until the end of each protocol. Afterwards, he will sit for 60 minutes of initial rest and HR, Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP), oxygen saturation (SpO2) and Heart Rate Variability (HRV) will be measured. After these measurements, volunteers will go to the second phase:

Placebo protocol (PP): consisting of the prior consumption of 3g of placebo (starch) and subsequently resting for 60 minutes, sitting, then a submaximal exercise test on an ergometric treadmill or;

Arginine (PA) experimental protocol: in this stage, volunteers will perform activities similar to the PC, but they previously consumed 3g of L-arginine 60 minutes before the submaximal test and then;

Perform physical exercise on a treadmill with a 1% incline for the first 3 minutes to warm up at a speed of 5km/h, followed by load increments of 1km/h every 2 minutes until reaching 80% of the maximum HR estimated by age (208-( 0.7*age) with the same inclination. At the end of the activity, you will remain lying down in a calm environment where HR, SBP, DBP, Spo2 and HRV will be monitored for another 20 minutes in the 1st, 3rd, 5th, 7th, 10th and 20th. minute.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged between 18 and 30 years, body mass index (BMI) between 18.5 and 29.9 kg/m2 and physically active according to the international physical activity questionnaire

Exclusion Criteria:

* Individuals who are sedentary and insufficiently active according to the IPAQ questionnaire, who present cardiorespiratory, neurological, renal, endocrine, metabolic, musculoskeletal disorders and other known or reported impairments that prevent the subject from performing the procedures, smokers, alcohol drinkers, users of medications that influence the autonomic nervous system and individuals with systolic pressure greater than 130 mmHg and diastolic pressure greater than 85 mmHg at rest

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Autonomic Nervous System | 10 minutes previous to exercise and 20 minutes after exercise.
  Heart Rate Variability

SECONDARY OUTCOMES:
Blood Pressure | 10 minutes previous to exercise and 20 minutes after exercise.
Heart Rate | 10 minutes previous to exercise and 20 minutes after exercise.
Oxygen Saturation | 10 minutes previous to exercise and 20 minutes after exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- UNESP, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No